CLINICAL TRIAL: NCT04673721
Title: PROSPective Evaluation of Fortified Eggs Related to Improvement in The Biomarker Profile for Your Health
Acronym: PROSPERITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eggland's Best (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: Pro00105996
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Hypercholesterolemia; Hyperlipidemia; Vitamin Deficiency; Obesity
Keywords: Fortified eggs; High cholesterol
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Avitaminosis; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fortified eggs + Intermittent fasting (Active Comparator): Consume at least 12 fortified eggs per week with 16-hour fast and then an 8-hour nutritional window.
  Interventions: Dietary Supplement: Fortified eggs; Behavioral: Intermittent fasting
- Non-egg supplemented diet + Intermittent fasting (Active Comparator): Maintain consumption of 2 or less eggs per week with 16-hour fast and then an 8-hour nutritional window.
  Interventions: Behavioral: Intermittent fasting; Dietary Supplement: Non-egg supplemented
- Fortified eggs + Usual care diet (Active Comparator): Consume at least 12 fortified eggs per week with consistency with current diet.
  Interventions: Dietary Supplement: Fortified eggs; Behavioral: Usual care diet
- Non-egg supplemented diet + Usual care diet (Placebo Comparator): Maintain consumption of 2 or less eggs per week with consistency with current diet.
  Interventions: Dietary Supplement: Non-egg supplemented; Behavioral: Usual care diet

INTERVENTIONS:
Dietary Supplement: Fortified eggs — Average 12 eggs consumed per week
  Arms: Fortified eggs + Intermittent fasting; Fortified eggs + Usual care diet
Behavioral: Intermittent fasting — 16-hour fast and then an 8-hour nutritional window with aim for energy needs to be consumed during an 8 hour eating window (e.g., 11 am - 7 pm) with fasting for 16 hours (e.g., 7 pm - 11 am the next day).
  Arms: Fortified eggs + Intermittent fasting; Non-egg supplemented diet + Intermittent fasting
Dietary Supplement: Non-egg supplemented — 2 or less eggs consumed per week
  Arms: Non-egg supplemented diet + Intermittent fasting; Non-egg supplemented diet + Usual care diet
Behavioral: Usual care diet — Consistency with current diet without consideration of intermittent fasting
  Arms: Fortified eggs + Usual care diet; Non-egg supplemented diet + Usual care diet

SUMMARY:
The objective of the study is to assess the effect of fortified eggs (compared to a non-egg supplemented diet) and intermittent fasting (IF) (compared to a usual care diet) on biomarker profile at 4 months. This will be a 140-participant, 2x2 factorial, randomized clinical trial comparing fortified eggs vs. a non-egg supplemented diet and IF vs. usual care diet through 4 months. Participants will be randomized 1:1:1:1 to the four treatment groups. Participants will have in-person follow-up visits at 1- and 4- months (inclusive of laboratory assessments) in addition to telephone calls at months 2 and 3. A subset of patients (~24 in each egg randomized strata) will undergo microbiome assessment at baseline and at 4 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years of age AND
* At least one of the following two criteria:

  * Prior cardiovascular event (myocardial infarction, coronary revascularization or ischemic stroke) OR
  * 2 cardiovascular risk factors including: 1) Diabetes mellitus (Defined as taking a medication for diabetes OR HgbA1c ≥6.5% within the prior 18 months; patients with diabetes may be treated with medications that are not associated with hypoglycemia such as metformin, thiazolidinediones (TZDs), glucagon-like peptide-1 receptor agonists (GLP-1 RAs), sodium glucose co-transporter 2 (SGLT2) inhibitors and/or dipeptidyl peptidase-4 (DPP-4) inhibitors, 2) Body mass index (BMI) ≥ 30 kg/m2, 3) Hypertension (Defined as taking blood pressure lowering medications OR systolic BP > 140mmHg at screening OR diastolic BP > 90mmHg at screening), 4) Dyslipidemia (Defined as taking lipid lowering medication OR LDL ≥130 OR HDL <50 for women OR HDL <40 for men OR triglycerides ≥150), or 5) Chronic kidney disease (Defined as eGFR <60 on most recent laboratory assessment within prior 18 months)
* Signed informed consent

Exclusion Criteria:

* Known allergy or intolerance to eggs
* Patients with diabetes who are on insulin or insulin secretagogues (e.g., sulfonylureas and meglitinides)
* Recent cardiovascular event (MI, stroke, HF hospitalization) within the past 30 days
* Planned initiation/change in lipid therapy within the next 4 months
* Current daily use of any supplements or multivitamins containing Vitamin B2 (riboflavin), Vitamin B12, Vitamin D, Vitamin E, or selenium or planned initiation within the next 4 months (current users need a 1-month washout period off supplement prior to eligibility)
* Inability or unwillingness to comply with the study requirements
* History of heart transplant or left ventricular assist device
* Pregnant or nursing women
* Malignancy or other non-cardiac condition limiting life expectancy to <4 months
* Consumption of > 2 eggs per week (this does not include eggs contained within other foods)
* Ongoing or recent (prior 30 days) participation in another interventional study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Change in LDL-cholesterol | Baseline, 4 months
Change in HDL-cholesterol | Baseline, 4 months

SECONDARY OUTCOMES:
Change in total cholesterol | Baseline, 4 months
Change in triglycerides | Baseline, 4 months
Change in NMP LipoProfile | Baseline, 4 months
Change in lipoprotein subfractionation | Baseline, 4 months
Change in apolipoprotein B | Baseline, 4 months
Change in fatty acid profile | Baseline, 4 months
Change in Vitamin B2 level | Baseline, 4 months
Change in Vitamin B12 level | Baseline, 4 months
Change in Vitamin D level | Baseline, 4 months
Change in Vitamin E level | Baseline, 4 months
Change in selenium level | Baseline, 4 months
Change in high-sensitivity troponin (hsTroponin) | Baseline, 4 months
Change in high-sensitivity c-reactive protein (hsCRP) | Baseline, 4 months
Change in hemoglobin A1c (HbA1c) | Baseline, 4 months
Change in insulin resistance score (LP-IR) | Baseline, 4 months

OTHER OUTCOMES:
Change in weight | Baseline, 4 months
Change in blood pressure | Baseline, 4 months
  Both systolic and diastolic blood pressure will be assessed
Change in Dietary intake (2005-Block Questionnaire) | Baseline, 4 months
Change in microbiome profile | Baseline through 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mentz, MD, FACC, FAHA, FHFSA, Principal Investigator — Duke Cardiovascular Disease Fellowship
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nouhravesh N, Harrington J, Aberle LH, Green CL, Voss K, Holdsworth D, Misialek K, Slaugh BT, Wieand M, Yancy WS Jr, Pagidipati N, Mentz RJ. Effects of fortified eggs and time-restricted eating on cardiometabolic health: The prosperity trial. Am Heart J. 2025 Jan;279:27-39. doi: 10.1016/j.ahj.2024.10.005. Epub 2024 Oct 15. PMID 39414223